CLINICAL TRIAL: NCT01225094
Title: Curcumin to Prevent Perioperative Complications After Elective Abdominal Aortic Aneurysm Repair: a Randomized Controlled Trial
Brief Title: Curcumin to Prevent Complications After Elective Abdominal Aortic Aneurysm (AAA) Repair
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Amit Garg, Professor, Medicine, Epidemiology & Biostatistics, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16593
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Acute Kidney Injury; Abdominal Aortic Aneurysm
Keywords: AAA; abdominal aortic aneurysm; acute kidney injury; ischemia-reperfusion
MeSH Terms: conditions — Acute Kidney Injury; Aortic Aneurysm, Abdominal | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- curcumin (Experimental): Patients will take the study medication (500 mg x 4 capsules, twice daily [BID]) for two days leading up to repair, totaling 4000 mg per day. They will take a dose (2000 mg) the morning of repair, at the same time as regular medications not held for surgery. While they are on call to the operating room, they will take another dose of 2000 mg., and then another 2000 mg dose 6 hours after the repair. Final dose (2000 mg)is administered morning after repair.
  Interventions: Drug: curcumin
- placebo (Placebo Comparator): The placebo will look, smell, taste, and in every way be identical to the active drug. Patients will take the study medication in the exact same manner as the curcumin regimen.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: curcumin — Patients will take the study medication (500 mg x 4 capsules, twice daily [BID]) for two days leading up to repair, totaling 4000 mg per day. They will take a dose (2000 mg) the morning of repair, at the same time as regular medications not held for surgery. While they are on call to the operating room, they will take another dose of 2000 mg and then another 2000 mg dose 6 hours after the repair. Final dose is administered the morning after repair.
  Other Names: NHPID name: curcumin
  Arms: curcumin
Other: placebo — The placebo will look, smell, taste, and in every way be identical to the active drug. Patients will take the study medication in the exact same manner as the curcumin regimen.
  Other Names: No brand name applicable.
  Arms: placebo

SUMMARY:
The purpose of this program of research is to determine whether curcumin, a natural health product, can prevent acute kidney injury and other complications after elective AAA repair. If proven safe and effective, curcumin is an inexpensive intervention which can be readily applied to almost 50,000 AAA repairs performed worldwide each year. New knowledge about this intervention may also guide its use in other surgical and medical settings to prevent complications to the kidneys, heart and other organs.

DETAILED DESCRIPTION:
An abdominal aortic aneurysm (AAA) is a ballooning of the abdominal aorta, the major blood vessel of the body. AAA occurs in up to 2% of adults. Surgeons will plan an AAA repair when the aneurysm grows bigger than 5.5cm, because the AAA might burst without repair. Over 47,000 AAA repairs are performed each year. Despite the benefits of AAA repair there are risks, and the kidneys can be severely injured. We will test whether the natural health product curcumin has an effect on biomarkers of inflammation, kidney injury and heart injury from AAA repair. Curcumin appears to fight oxidation and inflammation, which are ways that the body can be injured by surgery. We will study 600 patients who have elective AAA repair. The patients will receive either curcumin or a matching placebo. We will recruit the 600 patients from 10 centres in Ontario. This study will help us determine whether curcumin exerts any biological effect on biomarkers and whether it is well tolerated. If there is evidence of beneficial effects in this 600 patient trial, this will justify a future larger trial to assess the effects of curcumin on outcomes most important to patients, families and their healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

* Elective repair of an AAA (excludes thoracic or thoracoabdominal aneurysms)
* 18 years of age or older
* Able to provide informed consent
* Has one or more of the following criteria at time of preoperative assessment:
* x Open repair OR
* x Endovascular repair with ≥ 1 of the following criteria:
* o diabetes mellitus treated with insulin or oral hypoglycemic agents
* o age > 70 years
* o pre-existing renal impairment (baseline serum creatinine level >177 μmol/L for men or >146 μmol/L for women)
* If diabetic, is able and willing to collect and record glucose levels at home

Exclusion Criteria:

* emergent or urgent repair (repair < 3 days from pre-admission visit; ruptured AAA)
* prior renal transplantation
* pregnant or breastfeeding
* active gastrointestinal reflux disease, gastrointestinal ulcers or hepatobiliary disease (including gallstones)
* has active liver disease
* evidence of AKI (> 50% increase in serum creatinine) in the 30 days prior to repair
* enrolled in another randomized controlled trial
* receipt of ≥ 1 dialysis treatment in the past week
* previous participation in this trial
* repair is scheduled > 90 days from date of informed consent
* unable to provide written consent
* allergy(ies) to any member of the Zingiberaceae family: turmeric, ginger, curry, cumin, cardamom)
* allergy(ies) to ingredients of the study product or placebo: yellow or red food coloring, gelatin or cellulose
* have a history of major bleeding event in the previous 6 months
* bleeding disorders: a diagnosis of hemophilia, von Willebrand disease, platelets less than 70 for any reason
* history of hypoglycemia in the past 6 months: blood sugar less than or equal to 3.5 mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Urine IL-18 | Post op value
  We will examine the evidence of curcumin on biomarkers and whether it is well tolerated
NT-ProBNP | Change in post-operative minus pre-operative plasma NT-Pro BNP
hsCRP | Change in post-operative minus pre-operative plasma hsCRP
Serum creatinine | Change in peak post-operative serum creatinine (umol/L) in the 7 days following AAA repair minus pre-op value

SECONDARY OUTCOMES:
Binary measures of continuous biomarker outcomes | Continuous
  e.g acute kidney injury defined using accepted criteria
Safety outcomes | Peri-operative period
  Anemia, hypoglycemia, diarrhea, bleeding, peptic ulcer, nausea
Composite clinical outcomes adjudicated by investigators unaware of treatment outcomes | Within 30 days of AA repair
  New acute dialysis, myocardial infarction, receipt of coronary revascularization, sepsis, pneumonia, non-fatal cardiac arrest, stroke, deep vein thrombosis, pulmonary embolism, lower limb amputation, ischemic bowel, congestive heart failure, death

OTHER OUTCOMES:
Other outcome measures | Peri-operative period
  Study medication adherence, length of hospital stay, pain, blood pressure 3 hours after repair, urine output 3 hours after repair, other urine and blood biomarkers, tracer outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Amit X Garg, MD, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (10):
- Canada (10):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Sudbury Regional Hospital, Greater Sudbury, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Civic Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Garg AX, Devereaux PJ, Hill A, Sood M, Aggarwal B, Dubois L, Hiremath S, Guzman R, Iyer V, James M, McArthur E, Moist L, Ouellet G, Parikh CR, Schumann V, Sharan S, Thiessen-Philbrook H, Tobe S, Wald R, Walsh M, Weir M, Pannu N; Curcumin AAA AKI Investigators. Oral curcumin in elective abdominal aortic aneurysm repair: a multicentre randomized controlled trial. CMAJ. 2018 Oct 29;190(43):E1273-E1280. doi: 10.1503/cmaj.180510. PMID 30373740
- See also: Medline Plus related topics: Aneurysms Aortic Aneurysm — https://medlineplus.gov/aneurysms.html
- See also: Drug Information available for: Curcumin — http://druginfo.nlm.nih.gov/drugportal/name/Curcumin
- See also: U.S. FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks